CLINICAL TRIAL: NCT07100145
Title: Efficacy of Coconut Gel Compared to Corticosteroid Gel in the Management of Oral Lichen Planus (A Randomized Controlled Clinical Trial With Biochemical Analysis)
Brief Title: Efficacy of Coconut Gel Compared to Corticosteroid Gel in the Management of Oral Lichen Planus
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shahenda Mahmoud Farid Mahmoud, Assistant lecturer of oral medicine and periodontology department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-Rec IM012414
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; coconut oil; TNF-alpha; IL-10
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Coconut Oil; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical coconut gel (50%) (Experimental): topical coconut gel (50%) four times per day (after every meal and before going to bed) for eight weeks
  Interventions: Other: Coconut oil
- Topical corticosteroid (Active Comparator): topical corticosteroid (triamcinolone acetonide 0.1%) four times per day for eight weeks
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Other: Coconut oil — The composition per 100 g of virgin coconut oil 50% in oral mucoadhesive gel will be coconut oil (50 ml), tween 20 (surfactant-2.5 g) or span 60 (surfactant-2.5 g), Carbopol 940 (gelling agent-1 g), triethanolamine (viscous organic compound-0.2 g) and vanillin (0.001 g)
  Other Names: coconut gel
  Arms: Topical coconut gel (50%)
Drug: Triamcinolone Acetonide — topical corticosteroid
  Other Names: kenalog in orabase
  Arms: Topical corticosteroid

SUMMARY:
In oral lichen planus ,Tumor necrosis factor-alpha (TNF-α) has a role in the progression of the disease, enhancing CD8+ cytotoxic T cells and plays a role in the malignant transformation of the lesion. IL-10 is an anti-inflammatory cytokine that controls the disease and maintain homeoastasis. Treatment for OLP includes corticosteroids which is the gold standard, although they have considerable side effects. The use of herbal medicine as an alternative therapy seems promising. Coconut oil has anti-inflammatory, antioxidant, and immunomodulatory properties, no adverse effects, easily available, cost-effective and simply extracted.The aim of this randomized controlled clinical trial is to compare the therapeutic effects of topical 50% coconut mucobioadhesive gel versus topical corticosteroid gel in the management of symptomatic OLP clinically and using biochemical analysis

DETAILED DESCRIPTION:
Patients with symptomatic OLP will be recruited in the study. Group 1, containing 15 patients will receive topical coconut oil while Group 2 containing 15 patients will receive topical corticosteroid four times per day for a period of 8 weeks. Clinical assessment including clinical score, area of marker lesion and visual analogue scale will be compared between the two groups. Salivary samples from patients in the two groups will be collected at baseline and after 8 weeks to assess the level of TNF-α and IL-10 biochemically using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and histologically proven Bullous/erosive or atrophic forms of OLP.

Exclusion Criteria:

* lichenoid lesions.
* Presence of systemic conditions as; serious active or recurrent infections, malignancy, diabetes mellitus, hypertension, or significant heart, liver, or renal diseases.
* Smoking.
* Known hypersensitivity to the treatment drugs or any of the ingredients.
* Pregnancy or breast-feeding.
* History of previous treatments potentially effective on OLP such as antimalarial agents, retinoids, corticosteroids or immunosuppressive drugs in the last 2 weeks for topical medications, and 4 weeks for systemic medications prior to starting the study.
* Loss of pliability or flexibility in the tissues involved by the oral lesions of lichen planus.
* Histological signs of epithelial dysplasia or lichenoid lesions within the biopsied sites.
* Vulnerable groups (handicapped, orphans and prisoners).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical score | change from baseline two, four, eight and 12 weeks
  0: represented no lesion/normal mucosa
  1. mild white striae/no erythematous area
  2. white striae with atrophic area less than 1 cm2
  3. white striae with atrophic area more than 1 cm2
  4. white striae with erosive area less than 1 cm2
  5. white striae with erosive area more than 1 cm2

SECONDARY OUTCOMES:
salivary levels of Tumor Necrosis Factor-alpha (TNF-α) and Interleukin-10 (IL-10) | The Salivary Sample for each patient will be taken at baseline and after 2 months treatment period
  The mean concentration of TNF-α and IL-10 in whole saliva of patients with OLP lesions will be measured by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Nevine H Kheir El Din, Professor, Study Director — faculty of dentistry Ain Shams University

IPD SHARING:
Plan to Share IPD: No
Data is available upon reasonable request